CLINICAL TRIAL: NCT06009718
Title: A Deep-learning-based Multi-modal Phonocardiogram(PCG) and Electrocardiogram(ECG) Processing Framework for Screening Depressed Left Ventricular Ejection Fraction (dLVEF) Using a Wearable Cardiac Patch
Brief Title: Artificial Intelligence (AI) Analysis of Synchronized Phonocardiography (PCG) and Electrocardiogram(ECG)
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology Department, Chief Physician, Ruijin Hospital
Other Study IDs: RJH-PEG
Record Dates: First submitted 2023-07-06; First posted 2023-08-24 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
Keywords: Phonocardiography (PCG); Electrocardiogram (ECG); Heart Failure (HF); depressed left ventricular ejection fraction (dLVEF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Model training group: Compare the results of PCG and ECG with UCG, and conduct model training analysis
- Model validation group: Compare the results of PCG and ECG with UCG, and conduct model validation analysis

SUMMARY:
The diagnosis of depressed left ventricular ejection fraction (dLVEF) (EF<50%) depends on golden standard ultrasound cardiography (UCG). A wearable synchronized phonocardiography (PCG) and electrocardiogram (ECG) device can assist in the diagnosis of dLVEF, which can both expedite access to life-saving therapies and reduce the need for costly testing.

DETAILED DESCRIPTION:
The synchronized PCG and ECG is wirelessly paired with the WenXin Mobile application, allowing for simultaneous recording and visualization of PCG and ECG. These features uniquely enable this device to accumulate large sets of acoustic data on patients both with and without heart failure(HF).

This study is a Case-control study. In this study, the investigators seek to develop an artificial intelligence (AI) analysis system to identify dLVEF (EF<50%) by PCG and ECG. All adults (aged ≥18 years) planned for UCG were eligible to participate (inpatients and outpatients). Specifically, the investigators will attempt to develop machine learning algorithms to learn synchronized PCG and ECG of patients with dLVEF. Then we use these algorithms to identify dLVEF subjects. The investigators anticipate to demonstrate the wearable cardiac patch with synchronized PCG and ECG can reliably and accurately diagnose dLVEF in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at RuiJin hospital for UCG
* Signed dated informed consent
* Commit to follow the research procedures and cooperate in the implementation of the whole process research
* UCG has been completed
* Age ≥ 18
* At least 8 consecutive cycles of sinus rhythm can be recorded

Exclusion Criteria:

* Patients with pacemakers
* Complete left bundle branch block or block or QRS wave widening>120ms
* Left chest skin damaged or allergic to patch
* Refusal to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is one-center cohort study. Patients undergo echocardiogram at Ruijin Hospital.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Determination of Heart Failure Disease | one time assessment at baseline (approx. 5 minutes)
  Heart Failure Disease was determined by EMAT （millisecond, ms）calculate from synchronized PCG and ECG signals using an artificial intelligence (AI) guided model.

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, MD, PhD, Principal Investigator — Ruijin Hospital, Shanghai Jiaotong School of Medicine; Wenli Zhang, MD, Study Director — Ruijin Hospital, Shanghai Jiaotong School of Medicine; Bei Song, MD, Study Chair — Ruijin Hospital, Shanghai Jiaotong School of Medicine
Locations (3):
- China (3):
  - Ruijin Hospital, Shanghai Jiaotong School of Medicine, Shanghai
  - Shanghai Chest Hospital, Shanghai Jiao Tong University School Of Medicine, Shanghai
  - Shanghai East Hospital, Shanghai